CLINICAL TRIAL: NCT00341887
Title: PHIDISA I: A Prospective, Observational Cohort Study of HIV Infection (Both Treated and Untreated) and Risk-Related Co-Infections in the South African National Defence Force (SANDF)
Brief Title: Epidemiological Study of HIV in the South African National Defense Force
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904096; 04-I-N096
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-11-07

CONDITIONS: HIV
Keywords: Screening; AIDS; Antiretrovirals; Military; Force readiness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

SUMMARY:
This project, called PHIDISA I, will screen uniformed personnel of the South African National Defense Force (SANDF) and their registered family members for HIV, hepatitis B and C, gonorrhea, syphilis, and chlamydia to determine the incidence and prevalence of these sexually transmitted diseases. It will identify people who may be eligible to participate in clinical trials for preventing or treating HIV disease and will provide information that will be helpful in developing policy and better care for people affected with HIV and other diseases.

This project is part of the South Africa-U.S. PHIDISA Programme-a collaboration between the South African Military Health Service (SAMHS) of the SANDF, the U.S. Department of Defense, and the U.S. National Institutes of Health-to help prevent HIV transmission among South African military and civilian employees and their families.

Uniformed SANDF personnel or their family members who are eligible for health services from the SAMHS may enroll in the study. Participants visit the clinic every 6 months for up to 5 years for the following tests and procedures:

* Fill out a demographic information questionnaire
* Fill out a HIV risk assessment questionnaire
* Fill out a quality of life questionnaire
* Blood test
* Urine test
* Review of test results and counseling session with a doctor or nurse

Patients who test positive for HIV have a physical examination and additional blood draws.

...

DETAILED DESCRIPTION:
The South Africa - U.S. PHIDISA Project is a cooperative HIV/AIDS treatment research initiative established in 2003 for a likely duration of at least five years. It is an extension of the Masibambisane Programme, which is a cooperative initiative to help prevent the transmission of HIV/AIDS among South African military and civilian employees and their families. The PHIDISA Project is a collaboration between the South African Military Health Service of the South African National Defence Force (SANDF), the U.S. Department of Defence and the National Institutes of Health of the United States.

The PHIDISA Project has conducted clinical and operational research in HIV/AIDS in military and military-associated civilian populations. Scientists engaged in the research have been from South Africa, the United States and Australia and represent military and civilian medical, research and academic institutions. The project has established clinical research infrastructure within the SANDF and a network of its clinics, sick bays and hospitals. This has established important biomedical and public health research capacity that can be used in the future to address health issues of critical importance for military force preparedness.

An Executive Committee that includes South African and U.S. members manages the PHIDISA Project. An independent External Advisory Committee advises the project.

As a result of this project, information will be generated to assist SANDF in its future decisions about how best to manage the HIV/AIDS epidemic in military settings to assure SANDF combat readiness and to expand the wealth of knowledge regarding the best way to treat HIV infections. As a project complimentary to the Masibambisane Programme it also is anticipated that the PHIDISA Project will also contribute to the success of HIV transmission prevention activities in the military. The results of the PHIDISA Project also may contribute to HIV/AIDS clinical management, and related policy decisions, in the South African civilian sector.

ELIGIBILITY:
* INCLUSION CRITERIA:

Uniformed SANDF personnel or family members 14 years of age or older of SANDF personnel who are registered as eligible for health services from the SAMHS.

Able to provide written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8676 (Actual)
Dates: Start 2004-01-14; Study Completion 2012-11-07

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Polis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (5):
- South Africa (5):
  - Phalaborwa Sickbay, Phalaborwa, Limpopo
  - Umatata Sickbay, Eastern Cape
  - Area Military Health Unit Free State Poli-clinic, Free State
  - Mtubatuba Sickbay, Kwazulu-Natal
  - 2 Military Hospital, Western Cape

REFERENCES:
- [Background] Rabkin M, El-Sadr W, Katzenstein DA, Mukherjee J, Masur H, Mugyenyi P, Munderi P, Darbyshire J. Antiretroviral treatment in resource-poor settings: clinical research priorities. Lancet. 2002 Nov 9;360(9344):1503-5. doi: 10.1016/S0140-6736(02)11478-4. No abstract available. PMID 12433534
- [Background] Grosskurth H, Gray R, Hayes R, Mabey D, Wawer M. Control of sexually transmitted diseases for HIV-1 prevention: understanding the implications of the Mwanza and Rakai trials. Lancet. 2000 Jun 3;355(9219):1981-7. doi: 10.1016/S0140-6736(00)02336-9. PMID 10859054
- [Background] Mellors JW, Munoz A, Giorgi JV, Margolick JB, Tassoni CJ, Gupta P, Kingsley LA, Todd JA, Saah AJ, Detels R, Phair JP, Rinaldo CR Jr. Plasma viral load and CD4+ lymphocytes as prognostic markers of HIV-1 infection. Ann Intern Med. 1997 Jun 15;126(12):946-54. doi: 10.7326/0003-4819-126-12-199706150-00003. PMID 9182471